CLINICAL TRIAL: NCT06193915
Title: Ultrasound Guided Hematoma Block vs. Blind Hematoma Block in Distal Radius Fractures, a Randomized Controlled Trial
Brief Title: Ultrasound Guided Hematoma Block in Distal Radius Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Pieter Veenstra, Principal investigator, Frisius Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230041
Record Dates: First submitted 2023-09-21; First posted 2024-01-05 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Distal Radius Fractures; Fracture Dislocation; Dislocated Wrist; Dislocated Radius
Keywords: Distal radius fracture; Ultrasound; Hematoma block
MeSH Terms: conditions — Wrist Fractures; Fracture Dislocation

STUDY DESIGN:
Masking Description: Because treatment in both groups are different (one group with and one group without ultrasound) it's not possible to mask the treating physician for the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided hematoma block (Experimental): Patients in this group will receive ultrasound guided hematoma block before reduction of their dislocated distal radius fracture.
  Interventions: Device: Ultrasound guided hematoma block.
- Blind hematoma block (Active Comparator): Patients in this group will receive standard treatment; hematoma block with palpation of the fracture site (blind hematoma block)
  Interventions: Procedure: Blind hematoma block

INTERVENTIONS:
Device: Ultrasound guided hematoma block. — Patients with a dislocated fracture of the distal radius will receive ultrasound guided hematoma block with 10mL lidocaine 2% to get real-time guidance of the given anesthesia into the fracture site before closed reduction of a distal radius fracture.
  Arms: Ultrasound guided hematoma block
Procedure: Blind hematoma block — Patients with a distal radius fracture will receive standard treatment; hematoma block with 10mL 2% lidocaine performed with palpation of the fracture site (blind hematoma block) before closed reduction of dislocated distal radius fractures.
  Arms: Blind hematoma block

SUMMARY:
This study will investigate the effectiveness of analgesia of ultrasound hematoma block compared to 'blind' hematoma block in patients with dislocated distal radius fracture.

DETAILED DESCRIPTION:
Distal radius fractures represent one of the most common injuries in the Emergency Department (ED). Proper treatment especially for dislocated fractures can minimize the chance of residual injury. For closed reduction anesthesia is essential for safety, satisfaction and result. Different methods of regional anesthesia can be used but hematoma block (HB) is the technique most often used in EDs in the Netherlands and recommended by Dutch guidelines. In practice however a HB, does not always lead to adequate anesthesia, this might be because of poor infiltration into the fracture site. Ultrasound could additionally provide real-time guidance of injection into the fracture site, maximizing the analgesic effect of HB. In this study the effectiveness of analgesia of ultrasound HB will be compared to 'blind' HB in patients with a dislocated distal radius fracture.

Patients with a confirmed dislocated fracture of the distal radius requiring closed reduction will be randomized to either ultrasound guided hematoma block or normal 'blind' hematoma block. NRS-scores will be given before, during and after hematoma block and during and after reduction of the fracture. These scores will be the primary endpoint of this study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years
* Confirmed fracture of the distal radius requiring closed reduction, defined as any off the following items(7):

  * >10 degrees of dorsal angulation;
  * >20 degrees of volar angulation;
  * >2 mm step-off intra-articular;
  * >3 mm radial shortening;
  * >15 degrees radial inclination;
  * Translation and non-intact radio-carpal alignment in the lateral view
  * Significant translation in the posterior-anterior(PA)-view.

Exclusion Criteria:

* No informed consent can be given (cognitive impairment, severe dementia, no knowledge of Dutch language e.a.)
* Neurovascular compromise or open fractures requiring (immediate) surgery or reduction.
* First reduction already performed
* Multi-trauma patients requiring other urgent procedures/tests or with respiratory or hemodynamical compromise
* Pre-existent osteosynthesis material in situ in the affected arm
* Skin injury (with exception of minor abrasions), local infection or recent burns hindering or contra-indicating the use of ultrasound and ultrasound gel
* Allergy for local anesthetics

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of analgesia during closed reduction of a distal radius fracture | NRS before, during and after (10-15 min) injection of hematoma block, NRS-score during closed reduction and after closed reduction (5 min)
  Pain reduction will be measured on a Numeric Rating Scale( NRS-scale; 0-10) at different moments

SECONDARY OUTCOMES:
Number of participants in which hematoma was aspirated during hematoma block | During hematoma block
  Measure of correct position of hematoma block if there is aspiration of blood (yes/no)
Procedural time of the Hematoma block | Time from insertion of the needle until needle is withdrawn out of the patient (up to maximum of 30 min.)
  Time needed to perform HB (blind or ultrasound-guided; from moment of localization of the fracture until the moment the needle is out of the patient)
Procedural time of the reduction | From moment physician is ready to start the reduction until cast is applied (up to maximum of 30 min.)
  Time needed to perform reduction of the fracture
Satisfaction of the HB provided by physician performing the HB procedure | 10-15 minutes after hematoma block
  measured on a 5-points Likert-scale (Very satisfied, Somewhat satisfied, Neither satisfied nor dissatisfied, Somewhat dissatisfied or Very dissatisfied)
Satisfaction of reduction provided by physician performing reduction measured | 10-15 minutes after closed reduction
  measured on a 5-points Likert-scale (Very satisfied, Somewhat satisfied, Neither satisfied nor dissatisfied, Somewhat dissatisfied or Very dissatisfied)
Satisfaction of the patient for procedure and reduction | 10-15 minutes after closed reduction
  measured on a 5-points Likert-scale (Very satisfied, Somewhat satisfied, Neither satisfied nor dissatisfied, Somewhat dissatisfied or Very dissatisfied)
Satisfaction of the nurse for procedure and reduction | 10-15 minutes after closed reduction
  measured on a 5-points Likert-scale (Very satisfied, Somewhat satisfied, Neither satisfied nor dissatisfied, Somewhat dissatisfied or Very dissatisfied)
Number of reductions | (up to) 10-15 minutes after last closed reduction attempt
  Defined as attempt(s) to align fracture and application of cast
Years of experience of treating physician in performing HB. | (up to) 10-15 minutes after last closed reduction attempt
  Years of experience of treating physician in performing HB.
Years of experience of treating physician with use of ultrasound. | (up to) 10-15 minutes after last closed reduction attempt
  Years of experience of treating physician with use of ultrasound.
Number of patients in which palpation of an evident step-off near fracture site was felt | During performing hematoma block
  Before performing hematoma block performing physician will palpate if there is a clear step-off near the fracture site (important especially in blind hematoma group)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Veenstra, Principal Investigator — Medisch Centrum Leeuwarden
Locations (1):
- Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: No